CLINICAL TRIAL: NCT03658109
Title: Systemic Lidocaine Infusion or Quadratus Lumborum Block (in Addition to Intrathecal Morphine) Versus Intrathecal Morphine Alone as Part of a Gynecology-Oncology Surgery Early Recovery Protocol
Brief Title: Lidocaine Infusion or Quadratus Lumborum Block and Intrathecal Morphine, Versus Intrathecal Morphine Alone
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Recruitment challenges due to COVID-19
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Prentiss Lawson, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56789013
Record Dates: First submitted 2018-08-13; First posted 2018-09-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible patients will undergo current standard enhanced recovery protocol (ERP) gyn-oncology protocol. All patients will receive intrathecal morphine as part of the existing ERP. They will then be randomized to receive; either lidocaine infusion, regional anesthesia truncal block (quadratus lumborum block), or intrathecal morphine alone. Patients will be randomized into either lidocaine (group 1), QL block (group 2), or intrathecal opioid alone (group 3) groups. There will be blinding of the patient and personnel involved in data collection, and patients will undergo either a posterior QL block with local anesthetic (group 2) or simulated QL block (groups 1 and 3; subcutaneous local anesthetic only) pre-operatively. All patients will also undergo a loading dose of lidocaine (groups 1) or saline (group 2 and 3) followed by continuous lidocaine infusion in the lidocaine group (group 1). Primary and secondary endpoints will be measured post-operatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine Bolus Infusion (Active Comparator): Patients will also undergo a loading dose of lidocaine, followed by continuous lidocaine infusion in the lidocaine group.
  Patients will undergo an injection of intrathecal opioid medication (morphine) preoperatively.
  Patients will undergo a simulated QL block.
  Interventions: Drug: Lidocaine Bolus Infusion; Drug: Saline Bolus Infusion; Procedure: Simulated QL block
- QL Block & Saline Bolus Infusion (Active Comparator): Patients will undergo a posterior QL block.
  Patients will undergo an injection of intrathecal opioid medication (morphine) preoperatively.
  Patients will receive a saline bolus infusion.
  Interventions: Procedure: QL block
- Intrathecal Morphine Alone (No Intervention): Patients will undergo an injection of intrathecal opioid medication (morphine) preoperatively.
  Patients will undergo a simulated QL block.
  Patients will receive a saline bolus infusion.

INTERVENTIONS:
Drug: Lidocaine Bolus Infusion — Patients will undergo Lidocaine Bolus infusion.
  Other Names: Systemic Lidocaine Bolus Infusion
  Arms: Lidocaine Bolus Infusion
Procedure: QL block — Patients will undergo a posterior QL block pre-operatively
  Other Names: Posterior QL block
  Arms: QL Block & Saline Bolus Infusion
Drug: Saline Bolus Infusion — Patients will undergo Saline Bolus infusion.
  Other Names: Placebo Saline Bolus Infusion
  Arms: Lidocaine Bolus Infusion
Procedure: Simulated QL block — Patients will undergo a simulated posterior QL block pre-operatively.
  Other Names: Simulated posterior QL block pre-operatively
  Arms: Lidocaine Bolus Infusion

SUMMARY:
This study may provide evidence for whether or not systemic lidocaine infusion offers significant advantage over truncal regional blocks in gynecology oncology surgery patients in terms of post-operative analgesia, recovery, and safety profile. Further, it may show whether there is any increased efficacy of adding truncal regional block or systemic lidocaine versus intrathecal opioid administration alone.

DETAILED DESCRIPTION:
Systemic administration of intravenous lidocaine has a number of observed and theoretical advantages in the perioperative period. Systematic review of perioperative lidocaine infusions has shown a reduction in early post-operative pain scores in patients undergoing abdominal surgery, positive effects for GI recovery, reduction in post-operative opioid requirements, reduction in the incidence of post-operative nausea and vomiting, and decreased length of hospital stay. They have been shown to modulate the surgery-induced stress response in colorectal surgery and abdominal hysterectomy. Thoracic epidural analgesia was better as compared to intravenous lidocaine in a RCT of patients undergoing laparoscopic colorectal surgery as part of an enhanced recovery program, though there was similar impact on recovery of bowel function.

Truncal regional anesthesia has been utilized in open and closed abdominal operations with various levels of efficacy. A statistically significant, though marginal clinical analgesic benefit, by recorded opioid consumption, has been concluded by meta-analysis in patients undergoing abdominal laparotomy, laparoscopy, or cesarean delivery after US-guided TAP block. There was not found to be any additional benefit of TAP block in patients who received a spinal anesthetic that included a long-acting opioid. The interpretation of results was noted to be limited by the heterogeneity of the included studies and analysis, though. The conclusions of one study of open prostatectomy, as part of an ERP, was that neither systemic lidocaine nor TAP block improved post-operative analgesia. Both IV lidocaine and TAP block groups showed a reduction in post-operative opioid consumption, though to an insignificant degree. It was noted as a possibility that the other interventions as part of the ERP, such as scheduled administration of IV acetaminophen, could have resulted in the non-significant decrease in post-operative opioid requirement. A recent review of the use of TAP blocks in major gynecological, non-obstetric, surgery, including total abdominal hysterectomy, concluded that TAP blocks may contribute to early post-operative analgesia, with marginal additional benefit if multimodal analgesic regimens including NSAIDs and acetaminophen are added. It was hypothesized by the authors that some of the limited benefit might be due to the fact that US-guided TAP blocks are primarily useful for somatic pain, but that major gynecologic surgery has a large visceral pain component. There are limited randomized studies involving Quadratus Lumborum block (QL) at this time. QL block has shown improved analgesia in abdominal operations as compared to TAP block and is thought to have potentially greater relief of visceral pain. There is a case report of motor weakness following anterior, lateral QL block for gynecologic laparoscopy, thought to be related to spread of the block to affect the L2 dermatome on one side. It has not been determined if this is a common occurrence or may be affected by the type of QL block performed.

Prior to this study, truncal regional anesthesia was used in the UAB Gynecology-Oncology Surgery Enhanced Recovery Program as an analgesic alternative for those who were not good candidates for intrathecal opioid injection. A comparison of QL block versus systemic lidocaine infusion or whether either of these interventions has utility over intrathecal opioid administration alone has yet to be described.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing gynecologic-oncology surgery involving a mid-line laparotomy incision and as part of the local ERP, who are initially identified as an outpatient
* 18 years of age or older

Exclusion Criteria:

* Pregnancy,
* BMI>45,
* Age >70,
* Actual weight <65 kg
* Severe COPD
* Severe asthma
* Other severe respiratory disease (ILD, etc.)
* Local anesthetic allergy
* History of cardiac arrhythmia or heart block
* CHF
* Use of oral anti-arrhythmia agents or lidocaine analogues (i.e. mexiletine)
* Inability to be a candidate for intrathecal opioid injection based on medical history and provider judgement

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on biological gender identity.
Enrollment: 1 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
PACU Post-operative opioid consumption | From 0 to 12 hours post surgery
  Total opioid consumption (measured in oral morphine equivalents)

SECONDARY OUTCOMES:
Length of PACU admittance to time of readiness for discharge from PACU | Time of PACU admittance to the time of PACU readiness for discharge, generally not more than 12 hours
  This outcome measure will reflect the total amount of time required for the patient to be deemed suitable for discharge from the PACU, starting from the time of admittance to the PACU.
PACU Sedation Scores | From 0 to 12 hours post surgery
  This score will be collected using the modified Aldrete scale, every 15 minutes for the first hour of PACU stay, and once per hour for any additional hour(s) of PACU stay using a method consisting of: Consciousness = fully awake (2 points), arousable (1 point), not responding (0 points). This scale is used to determine a participant's state of arousal. The range of the scale is from 0-2, with zero being the most unresponsive and two being the most responsive.
Length of hospital stay | Time of admission until time of discharge, generally not over 1 week
Ambulation on POD 0 and POD1 | From 0 to 96 hours post surgery
  Number of minutes spent ambulating, per subject and/or nurse reporting
Return to bowel function | From 0 to 96 hours post surgery
  Return to bowel function (return of flatus, BM, ability to tolerate PO), per subject and/or nurse reporting
Total Opioid Dose Utilized During Surgery | From one hour before surgery start time to one hour after procedure stop time
  likely expressed as mcg of fentanyl but may be converted to morphine equivalent dose if multiple opioids are used
Presence or Absence of Patient Controlled Analgesia | From 0 to 96 hours post surgery
  Whether or not a PCA is needed for post-operative analgesia (Y/N - per usual documentation in the EMR.
Time to First Opioid Use | From 0 to 96 hours post surgery
  time from admission to the floor to administration of first opioid medication (per usual nursing documentation in the EMR).
Average PACU Pain Score | From 0 to 12 hours post surgery
  This outcome will be measured by taking the average of the numerical pain scale used to assess a patient's pain levels throughout their time in the PACU. The numerical pain scale has a range of 0 to 10, with 0 being no pain and 10 being very severe pain.
Post Operative Pain Scores | From 0 to 72 hours post surgery
  This outcome will be measured by taking the value of the numerical pain scale used to assess a patient's pain levels throughout their time in the hospital that is closest to each 4 hours after the time of the anesthesia documentation finish
Average PACU opioid consumption | From 0 to 12 hours post surgery
  Average total amount of opioids consumed in the PACU
Post-operative opioid consumption | From 0 to 72 hours post surgery
  Post-operative opioid consumption (measured in oral morphine equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: Prentiss Lawson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States